CLINICAL TRIAL: NCT02958228
Title: The Effect of Computerized Cognitive Training on Mood and Thinking Style Amongst Patients in Inpatient Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Simon Blackwell, Postdoctoral Research Assistant, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 325
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Depression; Anxiety; Anhedonia
Keywords: Positive Affect; Mental Imagery; Cognitive Bias Modification; Cognitive Control Training
MeSH Terms: conditions — Depression; Anxiety Disorders; Anhedonia | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Positive Mental Imagery Training (PMIT) (Experimental): Computerized Positive Mental Imagery Training (PMIT), a form of mental imagery-based cognitive bias modification adapted from previous experimental (e.g. Holmes, Lang, & Shah, 2009) and clinical (e.g. Blackwell & Holmes, 2010) work. The intervention consists of 8 sessions completed over a period of 2 weeks. The training takes place alongside participants' treatment as usual (TAU) in the inpatient setting.
  Interventions: Behavioral: Positive Mental Imagery Training (PMIT); Other: Treatment as Usual
- Cognitive Control Training (CCT) (Active Comparator): An adaptive Paced Auditory Serial Addition Task (PASAT), adapted from that applied in previous studies (e.g. Siegle et al., 2007; Hoorelbeke et al., 2015). The intervention consists of 8 sessions completed over a period of 2 weeks. The training takes place alongside participants' treatment as usual (TAU) in the inpatient setting.
  Interventions: Behavioral: Cognitive Control Training (CCT); Other: Treatment as Usual
- Treatment as Usual (Active Comparator): Participants will receive their treatment as usual (TAU) within the inpatient setting, which may include group/individual psychological therapy, a range of therapeutic activities, and pharmacological treatment.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Positive Mental Imagery Training (PMIT)
  Arms: Positive Mental Imagery Training (PMIT)
Behavioral: Cognitive Control Training (CCT)
  Arms: Cognitive Control Training (CCT)
Other: Treatment as Usual

SUMMARY:
The purpose of this randomized controlled trial is to establish feasibility and provide initial estimates of efficacy of two computerized cognitive training procedures (a form of Positive Mental Imagery Training, PMIT, and a form of Cognitive Control Training, CCT) delivered as adjuncts to treatment as usual (TAU) in inpatient mental health treatment settings.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* Sufficient German language skills
* Receiving treatment in a participating inpatient clinic during the timeframe of the study (i.e. they must be able to complete the training entirely within their admission).

Exclusion Criteria:

* Existence of a condition or circumstances that would interfere with completion of the study procedures (e.g. severe visual impairment, neurological problem, acute psychosis or substance withdrawal symptoms)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
21-item positive subscale from the extended Positive and Negative Affect Schedules | Post-intervention (2 weeks post-baseline)
  The Joviality, Self-Assurance, Attentiveness, and Serenity subscales of the extended PANAS (PANAS-X; Watson & Clark, 1994) will be administered, following previous experimental research examining the effect of positive mental imagery on state mood (e.g. Holmes, Lang, & Shah, 2009). Participants will be asked to rate the items according to how they have been feeling 'in the past week, that is, during the past seven days, including today'.

SECONDARY OUTCOMES:
21-item positive subscale from the extended Positive and Negative Affect Schedules | Baseline, Follow-up (2 weeks after the post-intervention assessment)
  The Joviality, Self-Assurance, Attentiveness, and Serenity subscales of the extended PANAS (PANAS-X; Watson & Clark, 1994) will be administered, following previous experimental research examining the effect of positive mental imagery on state mood (e.g. Holmes, Lang, & Shah, 2009). Participants will be asked to rate the items according to how they have been feeling 'in the past week, that is, during the past seven days, including today'.
Dimensional Anhedonia Rating Scale | Baseline, Post-intervention (2 weeks post-baseline), Follow-up (2 weeks after the post-intervention assessment)
  An extended 26-item version of the Dimensional Anhedonia Rating Scale (DARS; Rizvi et al., 2015) will be administered.
Quick Inventory of Depressive Symptomatology - Self Report | Baseline, Post-intervention (2 weeks post-baseline), Follow-up (2 weeks after the post-intervention assessment)
GAD-7 | Baseline, Post-intervention (2 weeks post-baseline), Follow-up (2 weeks after the post-intervention assessment)
Positive Mental Health Scale | Baseline, Post-intervention (2 weeks post-baseline), Follow-up (2 weeks after the post-intervention assessment)
Prospective Imagery Test | Baseline, Post-intervention (2 weeks post-baseline)
Scrambled Sentences Test (SST) | Baseline, Post-intervention (2 weeks post-baseline)
Implicit Associations Test (IAT) | Baseline, Post-intervention (2 weeks post-baseline)

OTHER OUTCOMES:
Self-report mood/cognitions over the previous day (Likert scales) | Baseline, up to 2 weeks post-baseline
  Ratings will be made up to 8 times over the two-week intervention period (between baseline and post-intervention)
State mood pre and post each training session (Likert scales) | Baseline, up to 2 weeks post-baseline
  Ratings of state mood will be made pre and post each session of PMIT or CCT by participants in the Positive Mental Imagery Training and Cognitive Control Training arms.
Credibility/Expectancy Questionnaire | Baseline
Feedback Questionnaire | Follow-up (2 weeks after the post-intervention assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Simon E Blackwell, DClinPsych, Principal Investigator — Ruhr University of Bochum; Jürgen Margraf, PhD, Study Chair — Ruhr University of Bochum
Locations (2):
- Germany (2):
  - Nexus-Klinik, Baden-Baden
  - St. Marien Hospital Eickel, Herne

IPD SHARING:
Plan to Share IPD: Yes
It is planned to make individual participant data available on publication of the associated study results, via a publicly-available data repository such as Open Science Framework. Data made available will be the research data reported in the publication, with the exception of any data that could compromise participant anonymity.

REFERENCES:
- [Derived] Blackwell SE, Westermann K, Woud ML, Cwik JC, Neher T, Graz C, Nyhuis PW, Margraf J. Computerized positive mental imagery training versus cognitive control training versus treatment as usual in inpatient mental health settings: study protocol for a randomized controlled feasibility trial. Pilot Feasibility Stud. 2018 Aug 4;4:133. doi: 10.1186/s40814-018-0325-1. eCollection 2018. PMID 30123524